CLINICAL TRIAL: NCT01411618
Title: Efficacy of Essential Oil Mouthwash With and Without Alcohol: a 3-Day Plaque Accumulation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: ENRICO MARCHETTI, University of L'Aquila
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 11/2010/SC
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2010-02

CONDITIONS: Gingivitis; Periodontitis
Keywords: Antiplaque agents; chemical plaque control; oral hygiene; essential oils; alcohol; mouthwash
MeSH Terms: conditions — Gingivitis; Periodontitis | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- free alcohol essential oil moutwash (Experimental)
  Interventions: Other: free alcohol essential oil mouthwash
- alcohol containing essential oil mouthwash (Active Comparator)
  Interventions: Other: free alcohol essential oil mouthwash

INTERVENTIONS:
Other: free alcohol essential oil mouthwash — All subjects were instructed to rinse twice a day, in the morning and in the evening, with 20 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.

SUMMARY:
The daily removal of supragingival dental plaque is a major factor in the prevention of caries, gingivitis and periodontitis. Proper control of bacterial plaque is obtained through the mechanical removal of the biofilm by the proper use of the toothbrush and floss. However, some studies have shown that the mean time of brushing tooth surfaces is less than that required to obtain a proper cleaning 1 and only 2-10% of the patients use dental floss regularly and effectively 2. In addition, it has been demonstrated that even after education and motivation of the patient to the proper use of toothbrush and floss, its compliance is reduced with time 3. The result is the persistence of plaque in some areas, particularly on the interproximal surfaces of teeth. Many studies have demonstrated the effectiveness and usefulness of antiseptic mouthwashes containing active ingredients such as chlorhexidine (CHX) and essential oils (EO) to prevent and control the formation of plaque and gingivitis, when used in addition to mechanical procedures 4-7. Chlorhexidine is still the gold standard for its antimicrobial action and high substantiveness, but side effects, such as pigmentation, taste alteration and the formation of supragingival calculus limit its continued use 8. Essential oil (EO) mouthwashes have been used for years as an adjunct to brushing in addressing oral hygiene. Their effectiveness in controlling plaque and gingivitis are well documented in literature 9-14. They kill microorganisms by destroying their cell walls and inhibiting their enzymatic activity 15,16. Furthermore, phenolic compounds like EOs are known to interfere with the inflammation process 17,18. The antibacterial action is particularly effective for the ability of the mouthwash with EOs to penetrate the biofilm 19-21. The traditional EO mouthwashes contain ethanol, a chemical used to dissolve numerous substances in mouthwashes, including CHX. The concentration of ethanol present in the mouthwash with EOs is more than 20%, sufficient to dissolve the EOs but not enough to carry out a direct antibacterial effect 22,23. Many aspects against the use of alcohol in mouthwashes, such as its effects on the surfaces of composite restorations 24 and its possible role in the formation of oropharyngeal cancer are being discussed 25,26. Although a direct correlation of the cause and effect between the occurrence of oropharyngeal cancer and the use of mouthwashes with alcohol 27, has not demonstrated so far, it is considered desirable to eliminate ethanol for use in daily mouthwash, bringing in search of new formulations. Recently, an EOs containing mouthwash without alcohol was introduced on the European market (Daycare, Curaden, Kriens, and Suisse). To our knowledge, to date there are no published data on the effectiveness of this antimicrobial product. The rinsing with this mouthwash can cause fewer side effects but, in contrast, it may be less effective.

The aim of this study was to evaluate the inhibitory properties of a new alcohol free EO containing mouthwash with respect to the traditional mouthwash containing 21.3% ethanol, through a standard 3-days plaque regrowth model.

ELIGIBILITY:
Inclusion Criteria:

* a dentition with ≥20 evaluable teeth (minimum of five teeth per quadrant),
* no oral lesions
* no severe periodontal problems (no probing depth ≥5 mm)
* no removable prostheses or orthodontic bands or appliances

Exclusion Criteria:

* allergies to several mouthwash components

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
difference between the two groups using the Plaque Index by Quigley and Hein modified by Turesky | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, Division of Periodontology, L’Aquila, AQ, Italy

REFERENCES:
- [Derived] Marchetti E, Mummolo S, Di Mattia J, Casalena F, Di Martino S, Mattei A, Marzo G. Efficacy of essential oil mouthwash with and without alcohol: a 3-day plaque accumulation model. Trials. 2011 Dec 15;12:262. doi: 10.1186/1745-6215-12-262. PMID 22171999